CLINICAL TRIAL: NCT03993184
Title: The Effects of Bikram (Hot) Yoga on Vascular Health in Hypertensive Adults
Brief Title: The Effects of Hot Yoga on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018381
Record Dates: First submitted 2018-03-06; First posted 2019-06-20 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2021-03

CONDITIONS: Hypertension; Elevated Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 90-minute Hot Yoga Classes (Experimental): This group will complete 3, 90-minute hot yoga classes weekly for 12 weeks.
  Interventions: Behavioral: Hot Yoga
- 60-minute Hot Yoga Classes (Experimental): This group will complete 3, 60-minute hot yoga classes weekly for 12 weeks.
  Interventions: Behavioral: Hot Yoga
- Control (No Intervention): This group will maintain their current physical activity for 12 weeks.

INTERVENTIONS:
Behavioral: Hot Yoga — Bikram or hot yoga is a standardized series of 26 postures with two breathing exercises. Classes will be performed at local yoga studios in Austin, Texas and participants will be required to sign in for each session. All participants will receive 12 weeks of free classes for their participation.
  Arms: 60-minute Hot Yoga Classes; 90-minute Hot Yoga Classes

SUMMARY:
This study will examine the effects of a 12 week hot yoga intervention on vascular health in adults between the ages of 20 and 65. The investigators are seeking individuals with slightly elevated blood pressure and stage I hypertension who are not currently taking blood pressure medications or exercising regularly. Participants will receive 12 weeks of free yoga for their participation.

DETAILED DESCRIPTION:
This study will examine the effects of a 12 week hot yoga intervention on vascular health by assessing changes of pre-intervention and post-intervention measurements in ambulatory blood pressure, endothelial function, and arterial stiffness in adults between the ages of 20 and 65. The investigators are seeking individuals with elevated blood pressure and stage I hypertension who are not currently taking blood pressure medications or exercising regularly. Participants will receive 12 weeks of free yoga for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Elevated blood pressure or stage I hypertension;
* sedentary (not currently exercising regularly);
* not currently taking blood pressure medications.

Exclusion Criteria:

* Pregnancy;
* renal disease;
* prior heart attack;
* known coronary artery disease;
* history of stroke,
* heart failure, cardiac arrhythmias or chronic obstructive pulmonary disease (COPD);
* recent chest pain;
* heat intolerance;
* body mass index of 40 or more.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Averages in ambulatory blood pressure and vascular function | 24 hours
  Blood pressure monitoring using an arm cuff for one full day before and after the intervention

SECONDARY OUTCOMES:
Perceived stress | 5 minutes
  "Perceived Stress Scale" questionnaire will be filled out by participant before and after the intervention in order to asses current perception of stress of daily living. 10 total questions, scaled from 0 to 4, 4 being the most often a participant felt stress and carries a weight of 5 and 0 holds a weight of 1. Question 4, 5, 7, and 8 have reversed values where 0 is the most heavily weighted and 4 is the least. The total is added up upon completion of each test and can be compared to before and after values.
Brachial artery endothelial function | 15 minutes
  Ultrasound imaging of the upper arm before and after 5 minutes of lower arm cuff inflation (this cuff similar to a blood pressure cuff but smaller) before and after the intervention. Arterial diameter images will be analyzed for baseline and post-cuff release diameters and flow-mediated dilation will be quantified as the percentage change in arterial diameter from baseline.
Arterial Stiffness | 10 minutes
  Tonometry readings of the carotid and femoral artery pulses assessing pulse wave velocity before and after the intervention. Pulse wave velocity will be determined by dividing the distance traveled in millimeters by the time delay between the initiations of the carotid and femoral pulse waveforms in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gonzales, Study Chair — Texas State University IRB
Locations (1):
- Texas State University, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: No